CLINICAL TRIAL: NCT01502683
Title: Operative Strategies to Reduce Cerebral Embolic Events During Coronary Artery Bypass Surgery
Brief Title: Stroke Study: Operative Strategies to Reduce Cerebral Embolic Events During Coronary Artery Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michael Halkos, Assistant Professor of Surgery, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00046608; 1K23HL105892-01A1 (NIH)
Record Dates: First submitted 2011-12-28; First posted 2012-01-02 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Stroke
Keywords: Stroke; neurocognitive dysfunction; cerebral embolic events
MeSH Terms: conditions — Stroke; Cognition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Off-pump No Clamp (Experimental): Off-pump coronary artery bypass patients randomized to no clamp for proximal anastomoses.
  Interventions: Procedure: No aortic clamping
- Off-pump Partial Occluding Clamp (Experimental): Off-pump coronary artery bypass patients randomized to partial occluding clamp for proximal anastomoses.
  Interventions: Procedure: partial occluding clamp
- On-pump Single Cross Clamp (Experimental): On-pump coronary artery bypass patients randomized to single cross clamp for cardioplegic arrest and proximal anastomoses.
  Interventions: Procedure: single cross clamp
- On-pump Double Clamp (Experimental): On-pump coronary artery bypass patients randomized to cross-clamp for cardioplegic arrest and partial-occluding clamp for proximal anastomoses. This strategy involves the application of two clamps.
  Interventions: Procedure: cross clamp and partial occluding clamp

INTERVENTIONS:
Procedure: No aortic clamping — No aortic clamp used in this group. The aortic clamp is a standard cardiac surgical instrument used during cardiac operations, not a specific device used for this study.
  Arms: Off-pump No Clamp
Procedure: partial occluding clamp — The partial-occluding clamp is a standardized instrument used during coronary artery bypass surgery, it is not a specific device for this study.
  Arms: Off-pump Partial Occluding Clamp
Procedure: single cross clamp — The proximal anastomoses performed under single clamp is an alternative method during coronary artery bypass surgery. The single clamp essentially means that whole operation is done using the cross clamp, which is a standard instrument during cardiac operations, not a specific device for this study.
  Arms: On-pump Single Cross Clamp
Procedure: cross clamp and partial occluding clamp — Both an aortic cross clamp and partial occluding clamp are used in this arm. Neither the cross clamp nor the partial clamp are specific devices for this study but are standard cardiac surgical instruments used during coronary artery bypass surgery and cardiac surgery.
  Arms: On-pump Double Clamp

SUMMARY:
One of the most devastating complications of coronary artery bypass surgery (CABG) is postoperative stroke. While there are multiple causes of stroke after CABG, particles generated during handling of the aorta is believed to account for most neurologic effects. Handling of the aorta during CABG occurs several times during the operation. One strategy to reduce aortic handling is to avoid cardiopulmonary bypass altogether by using off-pump techniques (OPCAB). Another method is to avoid the use of aortic clamps and/or to use devices that do not require aortic clamping. This study will test the hypothesis that an off-pump (OPCAB) approach and devices to perform clampless surgery will result in the least amount of aortic handling and therefore the lowest incidence and frequency of neurologic adverse events.

DETAILED DESCRIPTION:
One of the most devastating complications of coronary artery bypass surgery (CABG) is postoperative stroke. While the etiology of stroke after CABG is multifactorial, atheroemboli generated during aortic manipulation is believed to account for most cerebral embolic events. Manipulation of the aorta during CABG occurs during aortic cannulation, institution and maintenance of cardiopulmonary bypass, and during aortic clamping and unclamping with either a cross-clamp, partial-occluding clamp, or both. One operative strategy to minimize aortic manipulation is to avoid cardiopulmonary bypass altogether by using off-pump techniques (OPCAB). Another method is to avoid the use of aortic clamps and to construct proximal aortocoronary anastomoses with facilitating devices that do not require aortic clamping. The effect of these strategies on reducing cerebral embolic events and the underlying mechanism for this reduction are not well-defined.

This study will test the hypothesis that an off-pump (OPCAB) approach and facilitating devices to perform clampless proximal anastomoses will result in the least amount of aortic manipulation and therefore the lowest incidence and frequency of cerebral embolic events. The approach associated with the lowest incidence of TCD-detected cerebral embolic events will also result in the lowest incidence and severity of postoperative neurocognitive decline. Transcranial Doppler ultrasonography is an established method to detect cerebral embolic signals during cardiac surgery and will be utilized to detect cerebral embolic events during the operation. After an on- or off-pump strategy is selected, patients will be subsequently randomized to one of two clamping strategies. There will be 4 groups of patients: 1) OPCAB patients randomized to no clamping (facilitating device); 2) OPCAB patients randomized to partial clamping; 3) on-pump patients randomized to double clamping; and 4) on-pump patients randomized to a single clamp strategy.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* undergoing primary isolated coronary artery bypass surgery
* ability to sign informed consent

Exclusion Criteria:

* history of preoperative stroke
* reoperative cardiac surgery
* salvage or emergency CABG
* known left ventricular or left atrial thrombus
* concomitant valvular or aortic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2011-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Cerebral embolic events measured via transcranial doppler ultrasound | Intraoperative cerebral embolic events
  Cerebral embolic events measured via transcranial doppler ultrasound

SECONDARY OUTCOMES:
Neurocognitive dysfunction | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Halkos, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital Midtown, Atlanta, Georgia, United States